CLINICAL TRIAL: NCT07101237
Title: Integrative Multimodal Imaging and Multi-omics Profiling of HCC Heterogeneity: a Translational Exploratory Study Leveraging CEUS, Elastography, SMI, PAI, Multi-omics Analysis, and AI-driven Modeling to Advance Precision Diagnosis and Therapeutic Optimization
Brief Title: An Exploratory Study on Developing an Integrated Approach Combining Multimodal Imaging and Multi-omics Characterization of Tumor Heterogeneity for Precision Diagnosis and Treatment Optimization in Liver Cancer.
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Muti-omics liver cancer
Record Dates: First submitted 2025-07-21; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2024-12

CONDITIONS: Hepatocellular Carcinoma (HCC); Intrahepatic Cholangiocarcinoma (ICC); Primary Liver Cancer
Keywords: liver cancer; HCC; contrast-enhanced ultrasound (CEUS); elastography; superb microvascular imaging (SMI); photoacoustic imaging (PAI)
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma; Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Multi-modal ultrasonic imaging system for liver cancer — Conventional ultrasound, SMI, shear wave /strain elastography, and CEUS will be conducted for HCC/ICC patients. All above the imaging examinations will be conducted at 1/2/3/4/5/6, 9/12/15/18/21/24, and 30/36/42/48/54/60 months after the postoperative/post-conversion therapy.

SUMMARY:
Primary liver cancer, mainly including hepatocellular carcinoma (HCC) and intrahepatic cholangiocarcinoma (ICC), represents the third leading cause of cancer-related mortality. Enhancing the precision of liver cancer diagnosis and providing early therapeutic efficacy and prognostic evaluation during clinical decision-making hold significant clinical importance. Ultrasound is the preferred imaging modality for liver cancer screening. Contrast-enhanced ultrasound (CEUS) can dynamically visualize the microvascular perfusion of liver cancer lesions. Liver elastography has become a commonly used clinical assessment tool for cirrhosis. Photoacoustic imaging (PAI), an emerging non-invasive functional imaging technique, enables visualization of specific molecules through their spectroscopic characteristics at designated wavelengths.

The objectives of this study include: (1) Conducting an observational investigation combining CEUS, elastography, and superb microvascular imaging (SMI) to collect imaging data; (2) Preserving tumor specimens from participants to investigate heterogeneous protein characteristics of primary liver cancer organoids using PAI; (3) Analyzing peripheral venous blood samples to study transcriptomic profiles. Artificial intelligence (AI) technology will be employed to establish models integrating ultrasound radiomics with tumor multi-omics characteristics, aiming to provide novel strategies for precision diagnosis and treatment of liver cancer.

Key questions：(1) How to develop a multimodal imaging model combining CEUS, elastography, and SMI for predicting differentiation of liver cancer, microvascular invasion (MVI) and prognosis; (2) Whether PAI can identify heterogeneous proteins in liver cancer organoids through specific spectral recognition; (3) Whether AI can integrate multi-dimensional data to establish models based on ultrasound radiomics and multi-omics features.

DETAILED DESCRIPTION:
1. Research Background Primary liver cancer, predominantly comprising hepatocellular carcinoma (HCC) and intrahepatic cholangiocarcinoma (ICC), ranks as the third leading cause of cancer-related mortality. In China, approximately 70% of liver cancer patients are diagnosed at intermediate or advanced stages, where localized therapies such as surgery and ablation yield limited efficacy, and targeted therapies exhibit low overall response rates in advanced cases. This may be attributed to the heterogeneity of liver cancer, which manifests at multiple molecular levels-including genomic, transcriptomic, and metabolomic variations-both across individuals and within individual tumors. Such heterogeneity leads to divergent therapeutic responses and clinical outcomes among patients with identical pathological types and stages. Therefore, there is an urgent need to develop preoperative diagnostic methods capable of early assessment and prediction of tumor heterogeneity to guide precision clinical decision-making.

   Ultrasound is the preferred imaging modality for liver cancer screening due to its cost-effectiveness, safety and widespread clinical adoption. Contrast enhanced ultrasound (CEUS), the secondary guideline-recommended imaging technique for liver cancer diagnosis, offers economic and low-risk advantages compared to first-line recommendations like dynamic contrast-enhanced CT or MRI. Liver elastography has become a standard clinical tool for assessing cirrhosis. Photoacoustic imaging (PAI), an emerging non-invasive functional imaging technology, enables visualization of specific molecules based on their spectroscopic characteristics at designated wavelengths. Extensive studies have demonstrated the significant value of combined photoacoustic/ultrasound imaging in the diagnosis and prognostic evaluation of various cancers, including breast cancer and melanoma.

   This study aims to: (1) Conduct an observational investigation combining CEUS, elastography, and superb microvascular imaging (SMI) to collect imaging data; (2) Collect tumor specimens from participants for investigating heterogeneous protein characteristics in primary liver cancer organoids using PAI; (3) Analyze peripheral venous blood samples to study transcriptomic profiles. Artificial intelligence (AI) will be employed to establish prognostic models integrating ultrasound radiomics and tumor heterogeneity multi-omics features, providing novel insights for precision diagnosis and treatment of liver cancer.
2. Research workflow

   1. Construction of a diagnostic and prognostic model for liver cancer based on multimodal imaging Ultrasound examinations will be performed by sonographers with over five years of abdominal ultrasound experience. All the imaging data will be recorded.During the procedure, patients will assume a supine position with a left lateral decubitus position. Conventional ultrasound, SMI, shear wave /strain elastography, and CEUS will be conducted. Baseline data will be collected preoperatively, followed by postoperative/post-conversion therapy follow-ups at 1/2/3/4/5/6, 9/12/15/18/21/24, and 30/36/42/48/54/60 months to gather additional imaging and clinical data.
   2. Screening of prognosis-related heterogeneous multi-omics features and development of risk assessment models in HCC/ICC Peripheral venous blood (6-10 mL) will be collected from HCC/ICC patients. Whole blood and serum samples will be preserved, with 3 mL of whole blood and serum stored at -80°C. Another 3 mL of whole blood will be lysed in 9 mL TRIzol and stored at -80°C for multi-omics analysis. Tumor specimens will also be preserved for multi-omics studies and organoid-based heterogeneous protein characterization. Prognosis-associated transcriptomic and proteomic features will be screened based on patient outcomes, and prognostic risk models will be constructed by integrating these multi-omics profiles with clinical characteristics.
   3. Development of a predictive model integrating multimodal imaging and tumor heterogeneity multi-omics features via novel knowledge transfer and model training strategies First, transfer learning method will be applied to adapt basic perceptual capabilities from HCC/ICC multimodal imaging data. Furthermore, deep interactive fusion of radiomic features and tumor heterogeneity multi-omics data will be performed to establish predictive models for degree of HCC/ICC differentiation, MVI and prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 and ≤70 years;
2. Both sexes eligible;
3. Diagnosed with primary HCC or ICC;
4. Scheduled for surgical resection or conversion therapy;
5. Pathologically confirmed HCC/ICC via surgery or biopsy;
6. Posterior margin of the lesion ≤ 8 cm from the skin surface.

Exclusion Criteria:

1. Pregnancy, lactation, or planned pregnancy during the study period;
2. History of other malignancies;
3. Cardiac, pulmonary, cerebral, or renal insufficiency;
4. Lesion depth >8 cm from the skin surface on ultrasound;
5. Massive ascites;
6. Poor compliance (e.g., inability to hold breath during examination);
7. Allergy to ultrasound contrast agents.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with HCC and ICC who prepared for surgical resection or conversion therapy
Sampling Method: Non-Probability Sample
Enrollment: 308 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
tumor progression or follow-up failure. | From date of enrollment until the date of first documented tumor progression, assessed up to 5 years
  Tumor progression criteria:
  1. Target lesions: Based on the smallest sum of the longest diameters recorded in the study, progression is defined as: a) A ≥ 20% increase in the sum of the longest diameters of target lesions, with an absolute increase of at least 5 mm, or b) The appearance of new lesions.
  2. Non-target lesions: Clear progression of existing non-target lesions and/or the emergence of one or more new lesions.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China